CLINICAL TRIAL: NCT06670859
Title: The Effect of Mobilization Coverall Designed for Intensive Care Patients on Anxiety, Comfort, Physical Privacy and Satisfaction:Crossover Randomized Controlled Trial
Brief Title: The Effect of Mobilization Coverall on Anxiety, Comfort, Physical Privacy and Satisfaction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hatice AKKAYA, PhD Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dr-2024
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-10

CONDITIONS: Intensive Care Unit; Mobility; Patient
Keywords: Intensive Care Unit; Mobilization Coverall; Physical Privacy; Comfort; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention-Control: (Active Comparator): Intervention-Control: includes the group of patients who will perform their first mobilization with a mobilization coverall and their second mobilization with a traditional hospital gown.
  Interventions: Other: Intervention-Control:
- Control-Intervention: (Sham Comparator): Control-Intervention: includes the group of patients who will perform their first mobilization with a traditional hospital gown and their second mobilization with a mobilization coverall.
  Interventions: Other: Control-Intervention

INTERVENTIONS:
Other: Intervention-Control: — Patients will complete the STAI before the first mobilization after surgery and then the patients' pain status and the level of anxiety they feel about their physical privacy with the mobilization coverall they will wear during mobilization will be assessed with the VAS.Than,will be asked to perform 4 activities (putting on the coverall-mobilization-sitting in the wheelchair and moving-taking off the coverall) with the overall.Than,will be asked to evaluate the indicator level that they think the coverall they wear protects physical privacy and the levels of comfort and satisfaction they feel about the coverall with the VAS.During the next mobilization,patients will be asked to perform the same application protocol with a traditional hospital gown.Participants who have tried both clothing designs will be interviewed about their experiences using 'interview form' their satisfaction.Than interview,participants will have completed the study by filling out the QUEST 2.0.
  Other Names: Mobilization Coverall
  Arms: Intervention-Control:
Other: Control-Intervention — Patients will complete the STAI before the first mobilization after surgery and then the patients' pain status and the level of anxiety they feel about their physical privacy with the traditional hospital gown they will wear during mobilization will be assessed with the VAS.Than,will be asked to perform 4 activities (putting on the gown-mobilization-sitting in the wheelchair and moving-taking off the gown) with the gown.Than,will be asked to evaluate the indicator level that they think the gown they wear protects physical privacy, and the levels of comfort and satisfaction they feel about the gown with the VAS.During the next mobilization, patients will be asked to perform the same application protocol with the mobilization coverall.Participants who have tried both clothing designs will be interviewed about their experiences using 'interview form' their satisfaction.At the end of the interview, participants will have completed the study by filling out the QUEST 2.0.
  Other Names: Traditional Hospital Gown
  Arms: Control-Intervention:

SUMMARY:
This study is designed as crossover randomized controlled trial to examine the effect of a mobilization coverall designed for intensive care patients on anxiety, comfort, physical privacy and satisfaction.

DETAILED DESCRIPTION:
Patients receiving treatment in intensive care after surgical operation often experience a lack of privacy, comfort and control. One of the most important external factors affecting the experience of patients in the hospital is clothing. Hospital Gowns are made of clothes with special design and have a special place in the hospital experiences of patients during the perioperative period. Today, most hospital gowns consist of a single front panel, two back panels, sleeves and Two laces, and have a design with an opening in the back section. The design does not provide optimal functionality either for the patient wearing the hospital gown or for the medical personnel taking care of the patient. The current hospital gowns do not cover the body sufficiently, causing the patient to be embarrassed and dishonoring. Patients also express that the current apron lowers their self-esteem and makes them feel powerless and embarrassed. Failure to ensure the detection of drainage tubes causes patients to have difficulty during mobilization, causing drainage tubes to be held by medical personnel or the patient during mobilization. Additionally, in patient-focused qualitative studies in the literature, traditional hospital gowns worn by patients during mobilization cannot be tied or fully closed; It has been revealed that patients are more likely to want to stay in bed because of the concern that a part of their body will remain exposed or that their backrest will be exposed while walking. In this study, in order not to postpone mobilization, which has a positive effect on improving bowel functions, reducing the duration of intensive care and hospital stay, and increasing patient satisfaction, especially in the postoperative period; reducing anxiety regarding mobilization; A mobilization suit will be designed to protect the patient's physical privacy and increase his/her physical activity by ensuring his/her comfort during mobilization, and its effectiveness will be investigated.

The study will be conducted as a prospective crossover randomized controlled trial. After obtaining verbal and written consent from the participants before the study, the study will conduct with various data collection forms. These forms are; Individual Identification Form and Visual Analog Scale (VAS), Interview Form, Spielberger's State and Trait Anxiety Inventory (STAI), The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) will be used. Patients will randomize.

First Stage: Mobilization Coverall Design

The first stage of the study includes reviewing the studies in the literature on traditional hospital gowns used in the hospital and having the artistic and technical drawings of the mobilization suit designed by the researcher with the information obtained as a result of the observations of the researchers in line with their clinical experience drawn by the fashion design department in the city where the director works. Then, expert opinions will be obtained to determine the requirements and usage contexts of the mobilization suit design, produce design solutions, create a better design, improve the mobilization suit and determine the necessary changes through the visuals containing the front and back views of the artistic and technical drawings obtained.

Second Stage: Evaluating the Effectiveness of the Mobilization Coverall

The second stage of the study will conduct a crossover randomized controlled trial (RCT) to determine the effects of a mobilization coverall designed for intensive care patients on anxiety, comfort, physical privacy, and satisfaction.

Intervention-Control: includes the group of patients who will perform their first mobilization with a mobilization coverall and their second mobilization with a traditional hospital gown. Control-Intervention: includes the group of patients who will perform their first mobilization with a traditional hospital gown and their second mobilization with a mobilization gown.

ELIGIBILITY:
Inclusion Criteria:

* Being literate in Turkish
* Having undergone a surgical operation
* Presence of a urinary catheter after surgery
* Presence of Jackson-Pratt and/or Hemovac Drain after surgery
* Agreeing to participate in the study

Exclusion Criteria:

* Patients who cannot be mobilized after surgery
* Not completing any phase of the study
* Wanting to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety | It will be evaluated 5 minutes before clothing wear during
  Patients' anxiety levels will be measured with the State and Trait Anxiety Scale.
  Scale 1-20. account, state anxiety scaleen STAI-1 and subsequent 21-40. The questions consist of a total of 40 questions and two parts, including STAI-2, which measures trait anxiety. The constant production of anxiety requires how the individual usually expresses it. The emotions and behaviors expressed in trait anxiety behavior are, according to their frequency. The highest score that can be obtained from the scale is 80 and the lowest score is 20. A high score indicates high anxiety, and a low score indicates low anxiety. Additionally, anxiety level can be graded according to the score range: 0-19 points: No anxiety, 20-39 points: Mild anxiety, 40-59 points: Moderate anxiety, 60-79 points: Severe anxiety, 80 points: Severe anxiety (panic). It is evaluated as.
Change in comfort | It will be evaluated 5 minutes after completing the 4 specified activities (putting on the clothes-mobilization-sitting in the wheel chair and moving-taking off the clothes)
  The level of comfort they felt with the clothes they wore during mobilization.In this section, the degree of comfort level will increase or decrease.
  This situation will be evaluated with the Visual Analog Scale (VAS). VAS is a horizontal line of 100 mm in length. According to VAS, 0 mm is the lowest level and 100 mm is the highest level.
Change in protect their physical privacy | It will be evaluated 5 minutes after completing the 4 specified activities (putting on the clothes-mobilization-sitting in the wheel chair and moving-taking off the clothes)
  The level of protect their physical privacy they felt with the clothes they wore during mobilization.In this section, the degree of protect their physical privacy level will increase or decrease.
  This situation will be evaluated with the Visual Analog Scale (VAS). VAS is a horizontal line of 100 mm in length. According to VAS, 0 mm is the lowest level and 100 mm is the highest level.
Change in satisfaction | It will be evaluated 5 minutes after completing the 4 specified activities (putting on the clothes-mobilization-sitting in the wheel chair and moving-taking off the clothes)
  The level of satisfaction they felt with the clothes they wore during mobilization.In this section, the degree of satisfaction level will increase or decrease.
  This situation will be evaluated with the Visual Analog Scale (VAS). VAS is a horizontal line of 100 mm in length. According to VAS, 0 mm is the lowest level and 100 mm is the highest level.
satisfaction level for the designed mobilization coverall | It will be evaluated 30 minutes after the patients have experienced both clothing designs
  It will be used to evaluate users' satisfaction for the designed mobilization coverall. This situation will be evaluated with the the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0).The survey questions, consisting of a total of 12 questions, are answered on a 5-point Likert scale, with higher scores indicating higher satisfaction (1=not satisfied at all, 5=very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Ayhan, PhD, Study Director — University of Health Sciences Turkiye Gulhane Faculty of Nursing Ankara, Turkey
Locations (1):
- Kutahya City Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacofsky MC, Auran RL, Williams A, Mauro S, Sietsema D. Exposure-Related Anxiety and Improving Patient Satisfaction with Medical Undergarments During Surgery: A Randomized Controlled Trial. J Bone Joint Surg Am. 2022 Aug 3;104(15):1380-1385. doi: 10.2106/JBJS.22.00126. Epub 2022 Jun 20. PMID 35726887
- [Background] Morton L, Cogan N, Kornfalt S, Porter Z, Georgiadis E. Baring all: The impact of the hospital gown on patient well-being. Br J Health Psychol. 2020 Sep;25(3):452-473. doi: 10.1111/bjhp.12416. Epub 2020 Apr 20. PMID 32314508
- [Background] Syed S, Stilwell P, Chevrier J, Adair C, Markle G, Rockwood K. Comprehensive design considerations for a new hospital gown: a patient-oriented qualitative study. CMAJ Open. 2022 Dec 20;10(4):E1079-E1087. doi: 10.9778/cmajo.20210271. Print 2022 Oct-Dec. PMID 36735235
- [Background] -Koç, Z., Bulut, S., Karaman, H. "Nursing Care According to the Functional Health Patterns Model in a Patient Diagnosed with Adolescent Idiopathic Scoliosis: Case Report". Anatolian Journal of Nursing and Health Sciences, 2019, 22(4), 319-330.
- [Background] Frankel R, Peyser A, Farner K, Rabin JM. Healing by Leaps and Gowns: A Novel Patient Gowning System to the Rescue. J Patient Exp. 2021 Jul 21;8:23743735211033152. doi: 10.1177/23743735211033152. eCollection 2021. PMID 34368427
- [Background] -Cho, K., "Redesigning hospital gowns to enhance end users' satisfaction". Family and Consumer Sciences Research Journal, 2006, 34(4), 332-349.
- [Background] -Ağaç, S., Emiroğlu, S., "Design Application for the Improvement of Patient Gowns Used in Surgical Operations", International Journal of Cultural and Social Research, 2018, 4(Special Issue 3), 60-78.